CLINICAL TRIAL: NCT00345059
Title: Single Agent Chemotherapy With Weekly Docetaxel vs Combination Chemotherapy in Second-line Treatment of Advanced Non Small Cell Lung Cancer
Brief Title: The DISTAL-2 Study: Docetaxel Alone or in Combination in Second-line Treatment of Advanced Non Small-Cell Lung Cancer
Acronym: DISTAL-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow accrual
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISTAL-2
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: second line; monochemotherapy; combination chemotherapy; platinum refractory; previously treated
MeSH Terms: interventions — Docetaxel; Vinorelbine; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- docetaxel (Active Comparator): single agent docetaxel
  Interventions: Drug: docetaxel
- docetaxel + vinorelbine OR gemcitabine (Experimental): docetaxel in combination with either vinorelbine or with gemcitabine
  Interventions: Drug: docetaxel; Drug: vinorelbine; Drug: gemcitabine
- docetaxel + capecitabine (Experimental): docetaxel in combination with capecitabine
  Interventions: Drug: docetaxel; Drug: capecitabine

INTERVENTIONS:
Drug: docetaxel
Drug: vinorelbine
  Arms: docetaxel + vinorelbine OR gemcitabine
Drug: gemcitabine
  Arms: docetaxel + vinorelbine OR gemcitabine
Drug: capecitabine
  Arms: docetaxel + capecitabine

SUMMARY:
The purpose of this study is to compare the overall survival of patients with advanced non small cell lung cancer treated with docetaxel as single therapy versus docetaxel in combination with either gemcitabine or vinorelbine or in combination with capecitabine.

DETAILED DESCRIPTION:
This study is for patients with previously diagnosed advanced non small cell lung cancer (NSCLC, stage IIIb or IV) who had progression of their disease during or after first-line therapy containing platinum. Patients will be assigned to receive 6 cycles of therapy from one of four treatment regimens:

* docetaxel
* docetaxel + vinorelbine
* docetaxel + gemcitabine
* docetaxel + capecitabine

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18
* Histological diagnosis of non small-cell lung cancer (NSCLC)
* Stage IIIb or Stage IV disease (in IIIb, previous treatment with chemotherapy + radiotherapy, or metastatic supraclavicular lymph nodes or pleural effusion)
* Disease in progression
* Previous chemotherapy with platinum-derivative (and with > 21 days from last administration)

Exclusion Criteria:

* ECOG performance status > 2
* Age > 75 years
* History of malignant neoplasm within the previous 5 years (except for baso- or spino-cellular skin carcinoma and in-situ carcinoma of the uterine cervix, provided they are being adequately treated)
* Previous treatment with docetaxel
* Presence of symptomatic cerebral metastasis
* Neutrophils < 2.0 x 109/l, platelets < 100,000/l, hemoglobin > 10g/dl
* Bilirubin < 1.5 x the upper normal limit
* SGOT , SGPT, or bilirubin > 1.25 x the upper normal limits except in the presence of hepatic metastasis
* Creatinine >1.25 x the upper normal limit
* Any concomitant pathology that would, in the Investigator's opinion, contraindicate the use of the drugs in the protocol
* Inability to comply with follow up
* Pregnant or nursing females

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
overall survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hospital, Avellino, Italy; Division of Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D., Principal Investigator — Second University of Naples, Italy; Chair Medical Statistics
Locations (24):
- Italy (24):
  - Azienda Ospedaliera Giovanni Paolo II, Sciacca, AG
  - Azienda Ospedaliera S. Giuseppe Moscati, U.O. di Oncologia Medica, Monteforte Irpino, AV
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Università di Chieti, Chieti, CH
  - Ospedali Riuniti, Foggia, FG
  - Ospedale Umberto di Frosinone, Frosinone, FR
  - Ospedale di Gaeta, Gaeta, LT
  - Div. di Medicina Generale Osp. dei SS. Benedetto e Geltrude -Presidio Osp. Di Cuggiono - Az. Osp. Di Legnano, Cuggiono, MI
  - Ospedale Civile di Legnano, Legnano, MI
  - Ospedale S. Paolo, Milan, MI
  - Ospedale S. Gerado, Monza, MI
  - Azienda Ospedaliera Carlo Poma, Divisione di Oncologia ed Ematologia, Mantova, MN
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Azienda Ospedaliera V. Cervello, Palermo, PA
  - Ospedale Buccheri La Ferla - Fatebenefratelli, Palermo, PA
  - U.L.S.S. 15 Regione Veneto, Cittadella, PD
  - Istituto Oncologico Veneto, Padua, PD
  - Azienda Ospedaliera Universitaria Senese, Siena, SI
  - Ospedale E. Morelli, Sondalo, SO
  - Presidio Ospedaliaro Alto Gardo e Ledro, Arco, TN
  - Azienda Ospedaliera Di Busto Arsizio, Saronno, VA
  - Divisione di Oncologia Medica, U.S.L.L. 13, Noale, VE
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli

REFERENCES:
- [Result] Gebbia V, Morena R, Frontini L, Aitini E, Daniele B, Gamucci T, Di Maio M, Morabito A, Gallo C, Gridelli C. The DISTAL-2 phase III randomized trial of single agent weekly docetaxel (wD) vs wD plus gemcitabine (G) or vinorelbine (V) vs wD plus capecitabine (X) as second-line treatment of advanced non-small-cell lung cancer (NSCLC) patients (pts). J Clin Oncol 26: 2008 (May 20 suppl; abstr 19057)
- [Result] Gebbia V, Gridelli C, Verusio C, Frontini L, Aitini E, Daniele B, Gamucci T, Mancuso G, Di Maio M, Gallo C, Perrone F, Morabito A. Weekly docetaxel vs. docetaxel-based combination chemotherapy as second-line treatment of advanced non-small-cell lung cancer patients. The DISTAL-2 randomized trial. Lung Cancer. 2009 Feb;63(2):251-8. doi: 10.1016/j.lungcan.2008.05.027. Epub 2008 Jul 15. PMID 18632181